CLINICAL TRIAL: NCT00211640
Title: A Proactive Approach to the Identification and Treatment of Men With BPH Inthe Primary Care Setting
Brief Title: Identification and Treatment of Men With BPH in the Primary Care Setting
Status: Completed | Type: Observational
Sponsor: Mid Michigan Health Centers (Other)
Other Study IDs: MMHC001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-08

CONDITIONS: No Conditions for This Study. All Male Patients 18 Years of Age or Older Were Administered the LUTS, MSHQ, and Patient Demographics Questionnaire

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Male patients between the ages of 18 to 100 years of age who entered the Mid Michigan Health Center were administered a patient demographic questionnaire, a Lower Urinary Tract Symptom (LUTS) questionnaire, and the Men's Sexual Health Questionnaire (MSHQ) without exception. The purpose of this study was to better identify symptoms of benign prostatic hyperplasia (BPH) with the intent to prescribe better and more helpful treatment options for patients demonstrating these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All male patients between the ages of 18 to 100 years

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100

CONTACTS AND LOCATIONS:
Overall Officials: Matt T Rosenberg, M.D., Principal Investigator — Mid Michigan HC Partner
Locations (1):
- Mid Michigan Health Centers, Jackson, Michigan, United States